CLINICAL TRIAL: NCT00564759
Title: Phase I/II Gene Therapy Study for X-Linked Chronic Granulomatous Disease
Brief Title: Gene Therapy for Chronic Granulomatous Disease
Acronym: CGD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 58/59; DeReG 31; KSG 31
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Granulomatous Disease, Chronic
Keywords: CGD
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: retroviral SF71-gp91phox transduced CD34+ cells — autologous ex-vivo retroviral transduced (SF71-gp91phox) CD34+ cells

SUMMARY:
The aim of the study is to evaluate the side effects and risks after infusion of retroviral gene corrected autologous CD34+ cells of the peripheral blood of chemotherapy conditioned (busulphan)patients with chronic granulomatous disease (CGD). Also gene corrected and functional active granulocytes in the peripheral blood and the engraftment in the bone marrow of the patients will be monitored an documented.

ELIGIBILITY:
Inclusion Criteria:

* x-linked Chronic Granulomatous Disease
* history of life-threatening severe infections
* no HLA-matched related or non-related donor
* therapy resistent life threatening infections/organ dysfunction
* no other treatment options e.g. BMT

Exclusion Criteria:

* < 18 years of age
* HIV infection
* life expectancy > 2 years
* infections treatable by conventional therapy (antibiotics, allogeneic granulocytes)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
safety, toxicity and feasibility | 2 years

SECONDARY OUTCOMES:
Engraftment of gene corrected stem cells, functional reconstitution of respiratory burst, clinical benefit | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD, PhD, Principal Investigator — Goethe University
Locations (1):
- University Hospital, Hematology, Frankfurt, Germany

REFERENCES:
- [Result] Ott MG, Schmidt M, Schwarzwaelder K, Stein S, Siler U, Koehl U, Glimm H, Kuhlcke K, Schilz A, Kunkel H, Naundorf S, Brinkmann A, Deichmann A, Fischer M, Ball C, Pilz I, Dunbar C, Du Y, Jenkins NA, Copeland NG, Luthi U, Hassan M, Thrasher AJ, Hoelzer D, von Kalle C, Seger R, Grez M. Correction of X-linked chronic granulomatous disease by gene therapy, augmented by insertional activation of MDS1-EVI1, PRDM16 or SETBP1. Nat Med. 2006 Apr;12(4):401-9. doi: 10.1038/nm1393. Epub 2006 Apr 2. PMID 16582916